CLINICAL TRIAL: NCT03678051
Title: A Randomized Trial of CBT4CBT for Women in Residential Treatment for Substance Use Disorders
Brief Title: CBT4CBT for Women in Residential Treatment for Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20012674
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Substance Use Disorders; Drug Abuse; Drug Addiction; Substance Abuse; Drug Use Disorders; Drug Dependence; Substance Addiction
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): Standard of care
  Interventions: Behavioral: Treatment as Usual (TAU)
- TAU+CBT4CBT (Experimental): TAU with access to the CBT4CBT program
  Interventions: Behavioral: Treatment as Usual (TAU); Behavioral: TAU+CBT4CBT

INTERVENTIONS:
Behavioral: Treatment as Usual (TAU) — Standard of care residential treatment
Behavioral: TAU+CBT4CBT — 45-minute web-based modules covering core concepts to substance use treatment. The information is presented via graphics and voiceovers and key concepts are illustrated with brief videos depicting the material. Participants will be scheduled for a minimum of two sessions/week over the 3.5 weeks post-randomization (7 modules). These seven sessions will provide protected time to access the interventions, but the women will be able to access the modules and complete homework as much as they wish.
  Arms: TAU+CBT4CBT

SUMMARY:
This project examines computer-delivered cognitive-behavioral intervention (CBT4CBT) as an adjunct to residential treatment for women with substance use disorders (SUD). The project will conduct a 2-arm randomized clinical trial (RCT) comparing post-discharge relapse rates for treatment as usual (TAU) with access to the CBT4CBT program vs. TAU in a residential sample of women with SUDs.

DETAILED DESCRIPTION:
Women with substance use disorders face unique barriers to substance use treatment, and as a result, are less likely to seek treatment for substance use than their male counterparts. Women's residential treatment settings have been shown to have higher rates of treatment completion and better outcomes; however, relapse rates for substance use are high, with estimates ranging from 40-60%. Cognitive behavioral therapy (CBT) has been identified as an evidence-based treatment known to improve relapse rates by teaching clients how to recognize and respond to their cues for substance use. Women may particularly benefit from CBT, as their relapse risk factors include depression, interpersonal stress, and relationship conflict.

Despite the effectiveness of CBT, its dissemination is hindered due to limited availability of trained clinicians, cost, and limited resources. Computer-based training for cognitive behavioral therapy (CBT4CBT) offers an opportunity to improve the quality and reach of treatment services that is both feasible and cost-effective. Studies to date have demonstrated the utility of CBT4CBT in outpatient settings; however, it has not yet been evaluated as an adjunct to residential treatment for SUDs.

The specific aims are to: 1) Examine feasibility for use of CBT4CBT in a residential treatment program for women with SUDs; 2) Conduct a small RCT comparing TAU with access to the CBT4CBT program (CBT4CBT; intervention) vs. treatment as usual (TAU; control) using relapse rates and days of use as primary treatment outcomes; 3) Exploratory analyses will identify other correlates (e.g., coping strategies, depression) of relapse at 4 and 12 weeks post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Female
* Meet DSM-5 criteria for a SUD (current)
* Own a smartphone
* Can return to facility for the 4 and 12-week follow-up visits.

Exclusion Criteria:

* Pregnant
* Cognitive or psychiatric impairment
* Language barriers that preclude informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Any Relapse | 12-week follow-up period
  Percent of participants experiencing any relapse (yes/no), defined as any substance use (alcohol or other drugs) by self-report (smartphone or in person) and/or urine drug toxicology or Breathalyzer during 12-week follow-up period.
Days of Use | 12-week follow-up period
  Number of days of any substance use in 12 weeks post-discharge.

SECONDARY OUTCOMES:
Time to Relapse: | 12-week follow-up period
  Number of days post discharge to first use of any substance.

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis Pickens, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parlier-Ahmad AB, Kelpin S, Martin CE, Svikis DS. Baseline Characteristics and Postdischarge Outcomes by Medication for Opioid Use Disorder Status Among Women with Polysubstance Use in Residential Treatment. Womens Health Rep (New Rochelle). 2023 Dec 15;4(1):617-626. doi: 10.1089/whr.2023.0082. eCollection 2023. PMID 38145229